CLINICAL TRIAL: NCT02411825
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of Repeated Subcutaneous Doses of SAR425899 in Healthy Male Subjects and Overweight to Obese Patients With Type 2 Diabetes Mellitus
Brief Title: Multiple Ascending Dose Study in Healthy Male Subjects and Overweight to Obese Male and Female Type 2 Diabetes Mellitus (T2DM) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TDR13700; 2014-004216-10 (EudraCT Number); U1111-1163-1209 (Other: UTN)
Record Dates: First submitted 2015-03-24; First posted 2015-04-08 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SAR425899; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- SAR425899 (healthy subjects) (Experimental): Once daily SC doses of SAR425899
  Interventions: Drug: SAR425899
- Placebo (healthy subjects) (Placebo Comparator): Once daily SC doses of placebo
  Interventions: Drug: placebo
- SAR425899 (T2DM Patients) (Experimental): Once daily SC doses of SAR425899 and two up titration steps in each dose cohort with metformin as background therapy
  Interventions: Drug: SAR425899; Drug: metformin
- Placebo (T2DM Patients) (Placebo Comparator): Once daily SC doses of placebo and two up titration steps in each dose cohort with metformin as background therapy
  Interventions: Drug: placebo; Drug: metformin

INTERVENTIONS:
Drug: SAR425899 — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Arms: SAR425899 (T2DM Patients); SAR425899 (healthy subjects)
Drug: placebo — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Arms: Placebo (T2DM Patients); Placebo (healthy subjects)
Drug: metformin — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Placebo (T2DM Patients); SAR425899 (T2DM Patients)

SUMMARY:
Primary Objective:

To assess in healthy adult male subjects:

* The tolerability and safety of 21-day repeated subcutaneous (SC) doses of SAR425899 including two up titration steps.
* Pharmacokinetic (PK) parameters of SAR425899 after ascending repeated SC doses in plasma.
* Pharmacodynamic (PD) effects on fasting and postprandial plasma glucose, insulin, biomarkers of lipid metabolism and fibroblast growth factor 21 (FGF21).

To assess in overweight to obese T2DM mellitus patients:

* The tolerability and safety after 28-day repeated SC doses of SAR425899 including 2 up titration steps.
* PK parameters of SAR425899 after ascending repeated SC doses in plasma and urine.
* PD effects on fasting and postprandial plasma glucose, insulin, C-peptide, incretin panel (total and active ghrelin, total peptide YY [PYY], total and active glucagon-like peptide -1 [GLP-1], glucagon and total gastric inhibitory polypeptide-1 [GIP]), body weight, FGF21, biomarkers of lipid metabolism and HbA1c.

DETAILED DESCRIPTION:
The total study duration is approximately 10-15 weeks.

ELIGIBILITY:
Inclusion criteria:

Healthy subjects:

* Males, between 18 and 55 years of age, inclusive.
* Body mass index (BMI) between 20.0 and 30.0 kg/m^2, inclusive; body weight between 50.0 and 120.0 kg, inclusive.
* Certified as healthy by comprehensive clinical assessment (detailed medical history, complete physical examination). Comorbidities of higher weight (eg, mild impaired glucose tolerance, mild hypertension, mild hyperlipidemia) are permitted unless, per investigator, these conditions hamper participation.
* Normal vital signs after 10 minutes resting supine:
* 95 mmHg <systolic blood pressure (SBP) <150 mmHg.
* 45 mmHg <diastolic blood pressure (DBP) <100 mmHg.
* 50 bpm <heart rate (HR) <100 bpm.
* Standard 12-lead electrocardiogram (ECG) parameters after 10 minutes resting in supine position within; 120 ms <PR <220 ms, QRS <120 ms, QTc ≤430 ms, normal ECG.
* Normal 24-hour Holter electrocardiography at screening.
* Laboratory parameters within normal range; however serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless subject has Gilbert syndrome) should not exceed upper laboratory norm (ULN).

T2DM patients:

* Males and females, 18-70 years of age.
* Body weight 50.0-150.0 kg, BMI 28.0 - 42.0 kg/m^2.
* Diagnosis of T2DM for at least 1 year with stable metformin prior to inclusion; comorbidities related to T2DM but otherwise healthy.
* Normal vital signs supine:
* 95 mmHg < SBP <160 mmHg
* 45 mmHg < DBP <100 mmHg
* 50 bpm < HR <100 bpm
* Normal standard 12-lead ECG in supine position unless abnormality is clinically irrelevant.
* Laboratory parameters in normal range unless abnormality is clinically irrelevant or strongly associated with T2DM; total bilirubin not to exceed ULN.
* Fasting plasma glucose ≥90 mg/dL.
* HbA1c ≥6.5% and ≤8.5%.
* Females: Sterilization at least 3 months before inclusion or postmenopausal.

Both:

* Signed written informed consent.
* Not supervised/confined for legal or administrative reasons.
* Male subject with partner of childbearing potential (including lactating women) must use double contraception method.
* Male subject with pregnant partner must use a condom up to 2 months after last dosing.
* Male subject agreed not to donate sperm up to 2 months after last dosing.
* Not undergoing physical training program/planning changes in activity; not vegetarian or following special diet.

Exclusion criteria:

Healthy subjects:

* History of clinically relevant disease/signs of acute illness.
* History of drug hypersensitivity/allergic disease.
* Smoking more than 5 cigarettes/day.
* Any medication within 14 days before inclusion or within 5 times elimination/pharmacodynamic half-life of the medication and during study; vaccination within last 28 days, biologics given within 4 months before inclusion.

T2DM patients:

* History/presence of clinically relevant disease/signs of acute illness not related to patient's metabolic status.
* History/presence of drug hypersensitivity or allergic disease.
* Smoking more than 5 cigarettes per day.
* If female, pregnancy/breast-feeding.
* Any intake of medication during treatment period and within 21 days before first dosing or within 5 times half-life of the medication, except: metformin, standard antihypertensive treatment, statins, acetyl salicylic acid.
* Thyroid hormone replacement is allowed if dose was stable for 3 months prior to screening.
* Individual background therapy, considered necessary for the patient's welfare, that could not be discontinued for the duration of the study, may be given at the discretion of the Investigator, with a stable dose (when possible) and only if its intake is unlikely to interfere with the investigational product.
* Treated with sulphonyl-ureas up to 3 months, proton pump inhibitors up to 1 week prior to dosing.
* Vaccination within last 28 days, any biologics within 4 months before inclusion.
* Severe hypoglycemia resulting in seizure/unconsciousness/coma/hospitalization for diabetic ketoacidosis in last 3 months before screening.
* Persistent hyperglycemia not controlled by metformin/diet/exercise.
* Diabetic neuropathy, retinopathy, nephropathy or renal impairment.
* Hepatic impairment.
* Unstable hypo- or hyperthyroidism.

Both:

* Headaches/migraine.
* Recurrent nausea/vomiting.
* Blood donation within 1 month before inclusion.
* Symptomatic postural hypotension, irrespective of decrease in BP, or asymptomatic postural hypotension defined as decrease in SBP ≥20 mmHg within 3 minutes when changing from supine to standing.
* History/presence of drug or alcohol abuse.
* Positive result: hepatitis B surface antigen, anti-hepatitis C virus antibodies, anti-human immunodeficiency virus 1 and 2 antibodies.
* Any condition affecting gastric emptying or absorption from GI tract.
* Surgically treated obesity, bariatric surgery.
* Severe dyslipidemia with fasting triglycerides >450 mg/dL.
* History of pancreatitis or pancreatectomy.
* Amylase/lipase >3 ULN.
* History of thyroid cancer or a genetic condition that predisposes to thyroid cancer.
* Elevated basal calcitonin.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 28 to 35 days

SECONDARY OUTCOMES:
Changes in vital signs | 28 to 35 days
Changes in physical examination | 28 to 35 days
Changes in ECG | 28 to 35 days
Changes in clinical laboratory parameters (hematology) | 28 to 35 days
Changes in clinical laboratory parameters (biochemistry) | 28 to 35 days
Changes in body temperature | 28 to 35 days
Change from baseline in biomarkers (FGF21) | 28 to 35 days
Change from baseline in biomarkers (lipid biomarker) | 28 to 35 days
Change from baseline in biomarkers (incretins) | 28 to 35 days
Assessment of pharmacokinetic parameters in blood (AUC) | 28 to 35 days
Assessment of pharmacokinetic parameters in blood (Cmax) | 28 to 35 days
Assessment of pharmacokinetic parameters in blood (t1/2) | 28 to 35 days
Assessment of pharmacokinetic parameters in urine (Ae0-24) | 28 to 35 days
Assessment of pharmacokinetic parameters in urine (fe0-24) | 28 to 35 days
Change from baseline in Body weight | 28 to 35 days
Change from baseline in Fasting Blood Glucose | 28 to 35 days
Change from baseline in Postprandial Blood Glucose | 28 to 35 days
Change from baseline in postprandial Insulin | 28 to 35 days
Change from baseline in postprandial C-peptide profiles | 28 to 35 days
Change from baseline in HbA1c | 28 to 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Berlin, Germany

REFERENCES:
- [Derived] Visentin R, Schiavon M, Gobel B, Riz M, Cobelli C, Klabunde T, Dalla Man C. Dual glucagon-like peptide-1 receptor/glucagon receptor agonist SAR425899 improves beta-cell function in type 2 diabetes. Diabetes Obes Metab. 2020 Apr;22(4):640-647. doi: 10.1111/dom.13939. Epub 2019 Dec 22. PMID 31808298
- [Derived] Tillner J, Posch MG, Wagner F, Teichert L, Hijazi Y, Einig C, Keil S, Haack T, Wagner M, Bossart M, Larsen PJ. A novel dual glucagon-like peptide and glucagon receptor agonist SAR425899: Results of randomized, placebo-controlled first-in-human and first-in-patient trials. Diabetes Obes Metab. 2019 Jan;21(1):120-128. doi: 10.1111/dom.13494. Epub 2018 Sep 16. PMID 30091218